CLINICAL TRIAL: NCT04180046
Title: Glioblastoma Lines as the Disease Model
Brief Title: Utility of Primary Glioblastoma Cell Lines
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Antonella Arcella, Principal investigator, Neuromed IRCCS
Other Study IDs: NeuroPath_01
Record Dates: First submitted 2019-06-26; First posted 2019-11-27 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Tumor; Brain Tumor
Keywords: glioblastoma; cell; mutation
MeSH Terms: conditions — Neoplasms; Brain Neoplasms; Glioblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Representative biopsy specimens of the removed brain tumor will be sterilely removed and subjected to mechanical trituration and subsequently to enzymatic digestion with collagenase 1 and 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the characterization of human malignant glioma cell lines is described. After mechanical and enzymatic digestion of glioblastoma human biopsies from Neuromed IRCCS Neurosurgery patients, the investigators analyzed the established cell lines by immunohistochemistry. The investigators have already characterized 10 cell lines and results revealed that not all cell lines are positive for glial fibrillary acidic protein (GFAP), but only one was positive: the so-called COGI cell line. Moreover, the expression of Isocitrate Dehydrogenase 1(IDH1) and alpha thalassemia/mental retardation syndrome X-linked protein (ATRX) was investigated in all established cell lines. COGI cell line was also positive for IDH1R132 mutation and for ATRX. The results of characterization were summarized in table 1.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most aggressive type of brain tumor arising from glial cells accounting for 52% of all parenchymal brain cancer cases and 20% of all intracranial tumors. GBM has pronounced mitotic activity, substantial tendency toward neoangiogenesis (microvascular proliferation), necrosis, and high proliferative rates. Because of their intrinsic infiltrative nature, GBM has a highly aggressive malignant clinical course. The adjuvant chemo-radiotherapy (RT) with temozolomide (TMZ) after maximal safe resection remains the standard of care.

Brain cancer is a unique because of the "blood-brain barrier", which severely restricts the bloodstream of the brain. While the blood brain barrier (BBB) is great for protecting the brain from danger, when the brain has cancer cells, the BBB can be a problem. Therefore, it is important to find new drug targets. The mechanisms underlying radio- and chemo-resistance are poorly understood. Recent studies suggest that up-regulation of the molecular target of rapamycin (mTOR) plays a pivotal role in determining resistance to treatment. The upregulation of mTOR in GBM has been reported by multiple experimental and pathological findings. Moreover, the up-regulation of mTOR is also the key for cell growth and cell proliferation as demonstrated by in vivo studies. In fact, specific factors derived from brain endothelial cells maintain glioblastoma stem-like cell expansion through the mTOR pathway. The key to successful treatment of glioblastoma will be no doubt in the realization that this clinic is an entity in biologic terms, more than one disease, and is likely that specific targeted therapies will be effective in molecularly defined subsets. In this way, the molecular classification of these tumors will be defined in clinically relevant terms based on the identification of markers that define subsets and are predictive of response to promising agents. Additional investigations and identifications of new biomarkers will help to better define the clinical and biologic subtypes of glioblastoma and an improved disease control. In short, the brain tumor has peculiar ad personam mutations. This is why the investigators have decided to set up primary lines starting from the patient's biopsy.

Expected results of the scientific research project:

In the first instance, the primary outcome will be to establish cell cultures and stem cells that faithfully reproduce in vitro the physiology of the tumor maintaining the same characteristics of patient's neoplasm

1. Evaluate the effect of new target drugs on the proliferation of primary and continuous human glioblastoma cell lines by setting up growth curves and methyl thiazolyl tetrazolium (MTT) toxicity assays.
2. Screening of natural and synthetic drugs using patient-derived primary glioblastoma cell lines
3. Characterize the mechanisms and proteins involved in the apoptotic and / or autophagic pathway with immunohistochemistry and western blot assays in control and treated cells.
4. Validation of previously identified molecular targets in preclinical models of brain cancers. The investigators are able to identify novel molecular determinants that can be targeted by pharmacological intervention to decrease or block the tumor growth.

Materials and methods

Tumor Specimen Collection and Cryopreservation

Resection specimens of glioblastoma (GBM) tumors (n = 20) were received sterile and freshly from Neuromed Neurosurgery. Tumor tissue samples were snap frozen in liquid nitrogen and stored in the gas phase above liquid nitrogen. Additionally, tumor tissue cubes (3 × 3 × 3 mm) were frozen vitally. For this procedure, tumor pieces were cut with a sterile scalpel blade, and 4 tumor pieces were transferred into a sterile cryo-tube in 1.5 ml freezing medium (fetal calf serum containing 10% DMSO), sealed in a freezing container (Nalgene, Rochester , USA), and placed immediately at -80 ° C. Until thawing, tubes were kept at -80 ° C (for at maximum of 6 weeks) or, after overnight cooling, transferred to nitrogen tank (for longer storage periods).

Patient Cohort

Clinical samples from 5 patients with WHO grade IV GBM and 3 patient with a relapsed Astrocytoma, WHO grade III and one with oligodendroglioma grade III (Table 1) were collected from the Neurosurgery department at Neuromed IRCCS. Prior informed consent was obtained.

Tissue Culture and Cell Line Establishment

With written consent from patients and/or in accordance with institutional guidelines, immediately after the resection collect tumor samples (200-500 mg of tumor is recommended) into a tube containing cold sterile stem cell media without growth factors. Transport the specimen immediately to the tissue culture hood for processing.

For surgeries at a remote site, cut the tumor sample into smaller fragments and place into a tube containing cold sterile stem cell media without growth factors (keep on ice) for transportation. The tumor can be processed within 2-3 hours after the resection. Tumor specimens from a pre-clinical animal model of human GBM tumor can also be collected and processed in the same way.

In sterile BSL II laminar flow hood, place the tumor into a 35 mm petri dish with 3 mL of Hank's balanced salt solution (HBSS). Wash tumor specimen (2 to 3 times) by transferring them sequentially to new 35 mm dishes filled with 5 mL HBSS to remove blood and debris. Aspirate excessive HBSS from the dish. Immediately cut the tumor into small fragments and mince with a sterile scalpel blade into approximately 1 mm3 fragments. The best yield can be achieved when tumors are minced to very small pieces. Add 3 mL of enzymatic digestion mixture (collagenaseD/DNase 1) to the minced tissue and collect the minced tissue with 5 mL disposable pipet, pipetting up and down a few times. Then, transfer the tumor fragments into 30 mL of pre-warmed enzymatic digestion mixture.The final concentration of enzymes should be 1 mg collagenase D and 0.1 mg DNase I per milliliter of HBSS. After digestion tissue single cells were washed and plated . The cell lines were identified with the first letters of patient's name and surname.

Growth Kinetics

Cells (5×10^5 cells) were plated in 5 ml media in quintuplicate in T25 culture flasks per cell line and allowed to attach for 48 h; vital cells were assessed by trypan blue staining and one flask was counted every 24 h for five consecutive days using a Neubauer chamber.

O6-methylguanine-DNA-methyltransferase (MGMT) promoter methylation analysis

For analyzing the MGMT promoter concerning methylation the MethyLight method was applied. Briefly, genomic DNA (gDNA) was subject to bisulfite conversion using the Epitect Bisulfite Kit (Qiagen, Hilden, Germany) according to the manufacturer's recommendations. A primer/probe combination specific for methylated MGMT promoter sequence was used (forward: 5'-GCGTTTCGACGTTCGTAGGT-3'; reverse: 5'-CACTCTTCCGAAAACGAAACG-3'; probe: 5'-6FAM-CGCAAACGATACGCACCGCGA-TMR-3'), with SensiFast Probe Kit (Bioline, Luckenwalde, Germany). Cytosine-phosphate-guanosine (CpG) Methylase (SssI) treated DNA served as calibrator, as it is considered as fully methylated. The collagenase gene 2A1 (COL2A1), was used as endogenous control (forward: 5'-TCTAACAATTATAAACTCCAACCACCAA-3'; reverse: 5'-GGGAAGATGGGATAGAAGGGAATAT-3'; probe: 5'-6FAM-CCTTCATTCTAACCCAATACCTATCCCACCTCTAAA-TMR-3'). The percentage of methylated reference (PMR) value was calculated by dividing the MGMT/COL2A1 ratio of the sample by the MGMT/COL2A1 ratio of the SssI-treated DNA, and multiplying by 100. Samples with a PMR value >4 were considered as methylated. All reactions were performed in triplicate.

Mutation analyses

Samples underwent analyses for the following loci: IDH1 R132 (exon 4), IDH2 R172 (exon 4), B-Raf V600 (exon 15), K-Ras G12, G13 (exon 2) and Q61 (exon 3) and TP53 exons 5 to 8. The desired genomic regions were amplified by PCR using specific primers. The polymerase chain reaction (PCR) was performed using MyTaqHS polymerase (Bioline) according to the manufacturer's recommendations. The PCR reaction was controlled by agarose gel electrophoresis and 15 µl of the products were purified using 3 units of FAST AP™ Alkaline Phosphatase (Fermentas, St. Leon-Rot, Germany) and 30U of Exonuclease I (Fermentas) by incubation at 37°C for 15 min and subsequent heat inactivation at 85°C for 15 min.

Success Rates

The investigator assessed attachment and outgrowth rates of 2 consecutive WHO grade IV GBM tumor samples and two relapsed Astrocytoma, when prepared fresh directly after resection (culture #4). After fresh preparation, cells attached in 100% of the cases. The four most rapidly and stable outgrowing pairs of cell cultures were subsequently characterized in detail. In the following, stable outgrowing cultures (could be passaged >10 times) are termed cell lines. Cell lines derived from fresh material were marked with the initials of the patient's name and surname to ensure anonymity while respecting the patient's privacy.

Immunohistochemistry

Representative cell line of each tumour were stained by Immunohistochemistry for Ki67(proliferation index estimated as a (%) percentage of positive cells in a field of 100), IDH1, ATRX (markers of brain tumors) and GFAP (glial marker) (Ventana, Tucson, Ariz.) was performed automatically with a Nexes instrument (Ventana). Antibody detection was performed using a multilink streptavidin-biotin complex method, and antibodies were visualized by a diaminobenzidine chromagen method. Negative control samples were incubated with primary antibodies only.

Results

Table 1

Cell line Vimentin GFAP Atrx IDH1 MET

COGI + + + FE +

CL + + + - -

CG + FE + - +

PAP + + + + +

DNA + FE + - -

DRA + + + FE -

ZAR 67/19 + FE + - -

VEM + + + + +

DA + - + - +

IP + FE + - -

On these established cell cultures, new substances, including natural substances, will be tested and used as adjuvant substances for traditional therapy with Temodal. In this project the investigator intends to use coumaric acid.

1. Evaluate the effect of coumaric acid on the proliferation of human glioblastoma cells: primary and continuous lines;
2. Investigate the mechanisms triggered by coumaric acid in the neoplastic cell to block its growth. Analyze the expression of regulatory cell cycle proteins in human glioblastoma cells after treatment with coumaric acid at various concentrations.
3. Evaluate the growth of human glioblastoma cells in an animal model (naked CD1 mice inoculated with a continuous line of human glioblastoma U87MG cells) and after coumaric acid treatment.

ELIGIBILITY:
Inclusion Criteria:

• Patients with brain tumor: Glioblastoma (grade IV WHO)

Exclusion Criteria:

* Patients with other types of cancer
* Patients with brain tumor recurrence

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the study population is represented by patients with glioblastoma from NeuromedIRCCS Neurosurgery, the patients have no age limits
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Establishment of primary glioblastoma cell lines | 2 years
  Obtaining tumor biopsies to generate primary glioblastoma cell lines. Cells will also be used for phenotypic, genetic (IDH mutation and MGMT promoter methylation) and immunohistochemical characterization (e.g. glial markers GFAP, IDH1, P53, ATRX and proliferation marker Ki67), natural and synthetic drug screening in order to assess a dose-response correlation, or other molecular and cellular techniques.

CONTACTS AND LOCATIONS:
Overall Officials: antonietta Arcella, PhD, Principal Investigator — Neuromed IRCCS
Locations (1):
- Neuromed IRCCS, Pozzilli, IS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dolecek TA, Propp JM, Stroup NE, Kruchko C. CBTRUS statistical report: primary brain and central nervous system tumors diagnosed in the United States in 2005-2009. Neuro Oncol. 2012 Nov;14 Suppl 5(Suppl 5):v1-49. doi: 10.1093/neuonc/nos218. No abstract available. PMID 23095881
- [Background] Kleihues P, Louis DN, Scheithauer BW, Rorke LB, Reifenberger G, Burger PC, Cavenee WK. The WHO classification of tumors of the nervous system. J Neuropathol Exp Neurol. 2002 Mar;61(3):215-25; discussion 226-9. doi: 10.1093/jnen/61.3.215. PMID 11895036
- [Background] Diao W, Tong X, Yang C, Zhang F, Bao C, Chen H, Liu L, Li M, Ye F, Fan Q, Wang J, Ou-Yang ZC. Behaviors of Glioblastoma Cells in in Vitro Microenvironments. Sci Rep. 2019 Jan 14;9(1):85. doi: 10.1038/s41598-018-36347-7. PMID 30643153
- [Background] Stupp R, Weber DC. The role of radio- and chemotherapy in glioblastoma. Onkologie. 2005 Jun;28(6-7):315-7. doi: 10.1159/000085575. Epub 2005 Jun 2. No abstract available. PMID 15933418
- [Background] Arcella A, Oliva MA, Staffieri S, Aalberti S, Grillea G, Madonna M, Bartolo M, Pavone L, Giangaspero F, Cantore G, Frati A. In vitro and in vivo effect of human lactoferrin on glioblastoma growth. J Neurosurg. 2015 Oct;123(4):1026-35. doi: 10.3171/2014.12.JNS14512. Epub 2015 Jul 17. PMID 26186026
- [Background] Arcella A, Oliva MA, Sanchez M, Staffieri S, Esposito V, Giangaspero F, Cantore G. Effects of hispolon on glioblastoma cell growth. Environ Toxicol. 2017 Sep;32(9):2113-2123. doi: 10.1002/tox.22419. Epub 2017 Jun 15. PMID 28618133
- [Background] Arcella A, Oliva MA, Staffieri S, Sanchez M, Madonna M, Riozzi B, Esposito V, Giangaspero F, Frati L. Effects of aloe emodin on U87MG glioblastoma cell growth: In vitro and in vivo study. Environ Toxicol. 2018 Nov;33(11):1160-1167. doi: 10.1002/tox.22622. Epub 2018 Sep 15. PMID 30218594
- [Background] Zhuang W, Qin Z, Liang Z. The role of autophagy in sensitizing malignant glioma cells to radiation therapy. Acta Biochim Biophys Sin (Shanghai). 2009 May;41(5):341-51. doi: 10.1093/abbs/gmp028. PMID 19430698
- [Background] Galan-Moya EM, Le Guelte A, Lima Fernandes E, Thirant C, Dwyer J, Bidere N, Couraud PO, Scott MG, Junier MP, Chneiweiss H, Gavard J. Secreted factors from brain endothelial cells maintain glioblastoma stem-like cell expansion through the mTOR pathway. EMBO Rep. 2011 May;12(5):470-6. doi: 10.1038/embor.2011.39. Epub 2011 Apr 1. PMID 21460795
- [Background] Lefranc F, Facchini V, Kiss R. Proautophagic drugs: a novel means to combat apoptosis-resistant cancers, with a special emphasis on glioblastomas. Oncologist. 2007 Dec;12(12):1395-403. doi: 10.1634/theoncologist.12-12-1395. PMID 18165616
- [Background] Havik AB, Brandal P, Honne H, Dahlback HS, Scheie D, Hektoen M, Meling TR, Helseth E, Heim S, Lothe RA, Lind GE. MGMT promoter methylation in gliomas-assessment by pyrosequencing and quantitative methylation-specific PCR. J Transl Med. 2012 Mar 6;10:36. doi: 10.1186/1479-5876-10-36. PMID 22390413
- [Derived] Oliva MA, Staffieri S, Castaldo S, Giangaspero F, Esposito V, Arcella A. Characterization of primary glioma cell lines derived from the patients according to 2016 CNS tumour WHO classification and comparison with their parental tumours. J Neurooncol. 2021 Jan;151(2):123-133. doi: 10.1007/s11060-020-03673-8. Epub 2021 Jan 4. PMID 33398536